CLINICAL TRIAL: NCT05396729
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Sleep Quality in Healthy Volunteers on the Plateau
Brief Title: Acupoint Stimulation Improves Sleep on the Plateau
Acronym: ASSOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XJH-A-20220525
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Sleep Disorder
Keywords: transcutaneous electrical acupoint stimulation; plateau; sleep disorder; healthy volunteer
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The stimulator is put in an opaque box
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical acupoint stimulation (Experimental): Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given for 30 minutes
  Interventions: Device: transcutaneous electrical acupoint stimulation
- Control (No Intervention): Electrodes are placed at acupoints but no electrical stimulation is given

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given for 30 minutes, twice a day for 3 days.
  Other Names: TEAS
  Arms: transcutaneous electrical acupoint stimulation

SUMMARY:
Sleep disorder is common in people going to plateau. Acupuncture and related techniques could be used for treatment of sleep disorder. In this trial the effect of transcutaneous electrical acupoint stimulation on sleep disorder in people going to plateau will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years
* first time to the plateau (altitude ≥3000 meters)

Exclusion Criteria:

* those who live in area with altitude ≥2000 meters, or travel to plateau in the last half year
* history of insomnia
* patients with contraindication to transcutaneous electrical stimulation, including skin damage, infection or implantable electrical device
* difficulty in verbal communication
* history of taking medicine to improve sleep during the last 3 months
* regular daily intake of large dose of tea or coffee (>400 mg of caffeine)
* suspected or existed abuse of drug or alcohol
* disease that influence sleep such as chronic pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
total sleep time in 5 days | from arrived at plateau to 5 days after arrival, in a total of 5 days

SECONDARY OUTCOMES:
sleep latency on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
sleep efficiency on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
  sleep efficiency=total sleep time/total recording time
number of awake on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
Pittsburgh sleep quality index on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
Score of Cognition Assessment on the third day | from arrived at plateau to 5 days after arrival, in a total of 5 days
  cognition assessment is done using Rey Auditory Verbal Learning Test
lowest saturation of pulse oxygenation on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
highest systolic blood pressure on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days
highest heart rate on the fifth day | from arrived at plateau to 5 days after arrival, in a total of 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No